CLINICAL TRIAL: NCT05448014
Title: The Effects of a Self-compassion Therapist-led Online Group Treatment for Adolescents With Distress, Anxiety and Depression
Brief Title: Self-compassion Therapist-led Online Group Treatment for Adolescents With Distress, Anxiety, and Depression
Acronym: CUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Inga Dennhag, PhD, lecturer, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EtikDnr2021-04357CUST1
Record Dates: First submitted 2022-06-20; First posted 2022-07-07 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Distress, Emotional; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Study design: A two-arm (treatment group vs. control group) pilot randomized controlled trial will be carried out with 40 adolescents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CFT group intervention (Experimental): Compassion Focused Therapy in Group on the internet
  Interventions: Behavioral: Compassion focused group therapy online
- Control group (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: Compassion focused group therapy online — Seven sessions of therapist-led online compassion-focused therapy in groups of 4-8 adolescents with mild to moderate symptoms of distress, anxiety, or depression. Trained therapists administer the CFT program in face-to-face meetings.
  Arms: CFT group intervention

SUMMARY:
Background: Distress, anxiety and depression are highly prevalent in school health care or primary care. Many of these conditions remain undiscovered and/or untreated. Compassion-focused therapy (CFT) is effective in the treatment of adults' distress and depression, and we will now evaluate the preliminary effect of a brief therapist-led online group CFT, feasibility, and acceptability in low-threshold distressed, anxious, and depressed adolescents. We use online group CFT to increase availability.

Purpose: The purpose of this study is to determine whether therapist-led online group CFT is feasible and acceptable for the treatment of depression in adolescents between 15 and 20 years of age, in Sweden. The preliminary effect will be calculated to examine if a larger experimental randomized controlled trial is justified.

Study design: A two-arm (treatment group vs. control group) pilot randomized controlled trial will be carried out with 40 adolescents. The effect, feasibility, and acceptability of the therapist-led online CFT in groups will be evaluated.

DETAILED DESCRIPTION:
Adolescence is a vulnerable period of growth and challenges, characterized by rapid physiological and emotional changes. All these changes happen at the same time as relationships expand. A developing self together with a pressure to "fit in" can lead to self-critic and distress. Without appropriate coping skills to manage these challenges, adolescents are more vulnerable to psychological problems. Distress, anxiety, and depression have also increased in the western world during the last years, and especially girls or young women are affected [1]. In addition, depressive disorders are the single largest contributor to global disability [2]. Adolescents-appropriate training in compassion may help adolescents successfully overcome the challenges in the future and help adolescents to take care of themselves.

Schools are not just about acquiring knowledge, they are playing a central role in cultivating necessary social, emotional, and ethical skills required to lead successful lives [3]. Recently, there has been a great interest in bringing mindfulness and compassion to educators and students.

The construct of compassion is defined by Paul Gilbert as a "sensitivity to suffering in self and others with a commitment to try to alleviate and prevent it" [4] and include compassion for oneself, compassion for others, and receiving compassion from others. Compassion strategies are core competencies in life, already taught by large religions as Christianity and Buddhism, but now in a modern version along with new neurobiological research and cognitive behavior therapy interventions. These skills or strategies can be taught, but have not yet been widely used in the contexts of adolescents [3].

Research supporting compassion focused therapy for depression Compassion focused therapy (CFT) was developed two decades ago and is a well-established talking therapy for depression and stress [5]. Compassion has a protective effect against depression and suicidality [6], in youth. Training in compassion is linked to well-being and perceived life satisfaction [7]. Meta-analytic findings of CFT on adults has recently showed moderate effects on stress, depression and anxiety [7]. Studies with adolescents are few. For example one small study [8] with 34 14-17 year old students found that a mindful self-compassion school program in six weeks was feasible and acceptable. The intervention group had significantly greater self-compassion and less depression than the waitlist control.

The CFT intervention Compassion Focused Training (CFT). The investigators have developed a new manual for CFT training with seven modules [9] including 1) what is compassion, 2) understanding myself, 3) life-compass, 4) self-compassion and my body, 5) feelings and compassion, 6) create balanced thoughts, and 7) imagination. CFT is an internet-delivered (zoom or teams) real time group training (for 15-20 years old adolescents), 1,5h, in seven weeks. The youth will receive a manual for practice. The investigators were inspired by Professor Paul Gilbert, Mary Welford, and Elaine Beaumont's approach [10], but the investigators have shortened and adapted Welford and Beaumont manual to Swedish context. In addition, the investigators are influenced by cognitive behavior principles. Functional analyses and thoughts records are for example, used. The intervention focuses on the present and not on processing memories. The intervention is made for primary care and school health. A psychotherapist/psychologist or social worker will lead the training.

Theory behind the studies Compassion focused therapy is a components-based approach that integrates evolutionary theory, neurobiology, attachment theory, affect theory, family theory, cognitive behavioral principles, and humanistic theory [4].

The originality of the project Even though CFT has shown good results for adults, there are only a few small CFT studies on adolescents. None of them provide internet-delivered therapy. Our short internet-delivered group intervention for youths will be unique and could possibly be a good preventive and healing intervention for schools. Primary care and school health care need more efficient methods for both preventing and treating distress, anxiety, and depression.

Many barriers limit treatment uptake, such as limited number of trained therapists, costs, compliance issues such as time off work, and transportation, associated with the need to attend weekly appointments [11]. Delivering CFT in groups on the internet may be an effective and acceptable alternative to therapist-delivered treatment in primary care and at school health care. especially for rural areas.

Internet delivered such as telehealth, minimize barriers in access to care and address health-care disparities. Furthermore, internet delivered therapy allows for culturally and linguistically competent providers to offer mental health services to adolescents who might not have access to such clinicians in their communities. Nevertheless, several challenges have been identified in the literature including technological issues (e.g., poor internet connection), privacy and confidentiality (e.g. finding a quiet and private location), and safety concerns [12,11]. More and better studies with more modern technology are needed to develop this further.

A quality assurance data plan has been written. The investigators will collect quantitative data through RED Cap, which is a web survey recommended by Umeå University [13]. Data from RED Cap is saved at Umeå University. Only anonymous data with code will be saved at RED Cap.

Multifactor authentication is required for logging in to "protective documents" at Umeå University, and also for RED Cap, Outlook, TEAMS and other O365 system. The investigators are storing sensitive data on Umeå University system for that: protective documents [14].

The investigators are following Swedish archive laws and are using a Umeå University system for that [15].

The investigators will do data checks to compare raw data over time if data quality is sustained. Check sum will be used for this.

A data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, and coding information if used and normal ranges if relevant, will be performed.

Standard Operating Procedures have been written to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

Data calculations To address outcomes, data will be screened for faulty values and dependent variables will be examined for normality.

Randomization exclude systematic differences between groups (CFT group (n=20) and control group (n=20, waitlist)) at baseline, so the investigators will only calculate differences in effect sizes (Hedge g and Cohens d) on baseline demographic and psychosocial variables.

Descriptive statistics will be calculated for CFT group and control group for pre- and post-intervention.

To assess whether the groups (CFT group and control group) differ on post values, the investigators will conduct three Ancovas controlling for baseline. Dependent variables: posttest of total score of Perceived Stress Scale, subscale anxiety and depression in Trauma Symptom Checklist for Children (TSCC). Independent variable: Groups (CFT group and control group). Controlling variables: pretest of total score of total score of Perceived Stress Scale, subscale anxiety and depression in Trauma Symptom Checklist for Children (TSCC).

The investigators will calculate Hedges' g scores for effect size of differences between groups. Hedges' g is similar to Cohen's d, but includes a correction factor for small samples. Nonsignificant differences with Hedges' g greater than .20 are considered meaningful and are interpreted according to convention: .20=small, .50=medium, .80=large.

Finally, several Ancovas will be conducted to examine whether differences between CFT group and control group changes in secondary outcomes were found.

The investigators will use an exploratory approach for not missing any changes and the significance level will be 0.05. This study will be underpowered, and the outcome will be used to calculate power for a larger RCT-study. The investigators will both calculate result for intention to treat and for those who have participated more than two times.

Within-participant change will be calculated with Reliable Change Index [16].

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of distress (≥ 22 in PSS) and/or
* Symptoms of anxiety (≥ 9 in subscale Anxiety in TSCC) and/or
* Symptoms of depression (≥ 10 in subscale Depression in TSCC)
* Adolescent giving informed consent
* Caregiver giving informed consent if needed
* Speaking Swedish
* Able to read and fill forms in Swedish without troubles
* At least one close and stable relationship with an adult
* Able to be in a group on the internet

Exclusion Criteria:

* Severe psychological problems that can be hindering for participation in a group treatment
* No close stable relationship with an adult
* Suicidal risk (4 or higher in item 12 in MADRS-Y, together with a clinical decision of active suicidal plans during the diagnostic screening interview)
* Bipolar Disorder
* Autism
* Anorexia Nervosa
* Current substance and alcohol dependence
* Current psychosis
* Current active psychotherapy
* Current deposit or withdrawal of antidepressant
* Prescribed medications for anxiety or depressive disorders do not exclude participants from the study, if the dosage had remained constant for at least one month.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inga Dennhag, PhD, Principal Investigator — Umeå University
Locations (1):
- Inga Dennhag, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. WHO (2019). Spotlight on adolescent health and well-being: Findings from the 2017/2018 health behaviour in school-aged children (HBSC) survey in Europe and Canada. In J. Inchley (Ed.), (Vol. 2).
- [Background] 2. World Health Organization (2017). Depression and other common mental disorders: Global health estimates. http://apps.who.int/iris/bitstream/handle/10665/254610/WHO-MSD-MER-2017.2-eng.pdf;jsessionid=5C6C365CE6CA46022D8AE57751200AE9?sequence=1.
- [Background] 3. Jazaieri, H. (2018). Compassionate education from preschool to graduate school: Bringing a culture of compassion into the classroom. Journal of Research in Innovative Teaching & Learning, 11(1), 22-66, doi:10.1108/JRIT-08-2017-0017.
- [Background] Gilbert P. The origins and nature of compassion focused therapy. Br J Clin Psychol. 2014 Mar;53(1):6-41. doi: 10.1111/bjc.12043. PMID 24588760
- [Background] 5. Gilbert, P. (2007). Psychotherapy and counselling for depression (3rd ed.). Los Angeles: SAGE.
- [Background] Zeller M, Yuval K, Nitzan-Assayag Y, Bernstein A. Self-compassion in recovery following potentially traumatic stress: longitudinal study of at-risk youth. J Abnorm Child Psychol. 2015 May;43(4):645-53. doi: 10.1007/s10802-014-9937-y. PMID 25234347
- [Background] Kirby JN, Tellegen CL, Steindl SR. A Meta-Analysis of Compassion-Based Interventions: Current State of Knowledge and Future Directions. Behav Ther. 2017 Nov;48(6):778-792. doi: 10.1016/j.beth.2017.06.003. Epub 2017 Jun 21. PMID 29029675
- [Background] Bluth K, Gaylord SA, Campo RA, Mullarkey MC, Hobbs L. Making Friends With Yourself: A Mixed Methods Pilot Study of a Mindful Self-Compassion Program for Adolescents. Mindfulness (N Y). 2016 Mar 1;7(2):479-492. doi: 10.1007/s12671-015-0476-6. Epub 2015 Dec 19. PMID 27110301
- [Background] 9. Dennhag, I. (2021). Att lära om Self-compassion [eng. To learn about Self-compassion]. (pp. 66). Umeå Universitet, Sweden: Clinical Science.
- [Background] 10. Welford, M., & Beaumont, E. (2020). The kindness workbook: Creative and compassionate ways to boost your wellbeing. London: Robinson Publishing.
- [Background] Simon N, Robertson L, Lewis C, Roberts NP, Bethell A, Dawson S, Bisson JI. Internet-based cognitive and behavioural therapies for post-traumatic stress disorder (PTSD) in adults. Cochrane Database Syst Rev. 2021 May 20;5(5):CD011710. doi: 10.1002/14651858.CD011710.pub3. PMID 34015141
- [Background] Stewart RW, Orengo-Aguayo RE, Cohen JA, Mannarino AP, de Arellano MA. A Pilot Study of Trauma-Focused Cognitive-Behavioral Therapy Delivered via Telehealth Technology. Child Maltreat. 2017 Nov;22(4):324-333. doi: 10.1177/1077559517725403. Epub 2017 Sep 4. PMID 28868894
- [Background] 13. Umeå University (2022). REDCap - data collection in research studies (In Swedish: REDCap - Datainsamling vid forskningsstudier). https://www.aurora.umu.se/stod-och-service/it-och-digitala-tjanster/samla-in-data/datainsamling-forskning/.
- [Background] 14. Umeå University (2022). Storing of files with high level of security (In Swedish: Lagra filer med högt skyddsvärde i Skyddade dokument). https://www.aurora.umu.se/stod-och-service/it-och-digitala-tjanster/dokument-fillagring/skyddade-dokument/. Accessed 2022-06-20.
- [Background] 15. Umeå University, & Clinical Science (2022). Research Archive Clinical Science (In Swedish Forskningsarkivet Klinisk Vetenskap). http://foark.klinvet.umu.se:5000/#/signin.
- [Background] 16. Blampied, N. M., Conference, N., & Wellington (2016). Reliable change & the reliable change index in the context of evidence-based practice: A tutorial review. https://ir.canterbury.ac.nz/handle/10092/13399
- [Derived] Vestin M, Wallin L, Naesstrom M, Blomqvist I, Svedin CG, Beaumont E, Jokinen J, Dennhag I. Internet-based group compassion-focused therapy for Swedish young people with stress, anxiety and depression: a pilot waitlist randomized controlled trial. Front Psychol. 2025 Apr 1;16:1547046. doi: 10.3389/fpsyg.2025.1547046. eCollection 2025. PMID 40236966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates: 1 June 2022- 1 dec 2023 Types of location: The current study was promoted to young people via social media, flyers, and direct outreach by project staff or personnel at schools and primary care health centers in northern Sweden.
Pre-assignment Details: N = 85 were assessed for eligibility. Excluded/not eligible (n = 43)
  1. Did not meet inclusion criteria (e.g. symptoms, age; n = 15)
  2. Severe condition (n = 6)
  3. Other treatment (n = 2)
  4. Drop out practical reasons (n = 10)
  5. Withdrew unknown reason (n = 10)
Groups:
- Control Group: Waiting list for Compassion Focused Therapy
Period: Overall Study
Arm/Group | CFT Group Intervention | Control Group
Started | 22 | 20
Completed | 18 | 13
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CFT Group Intervention | Control Group | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.1 (1.8) | 17.4 (1.7) | 17.2 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of participants
  Participants
    Female | 21 | 17 | 38
    Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 22 | 20 | 42
Perceived Stress Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The 10-item Perceived Stress Scale (PSS-10) measures perceived stress related to unpredictability, uncontrollability, and overload in daily life. Each item is rated on a 5-point scale from 0 (never) to 4 (very often), yielding a total score ranging from 0 to 40. Higher scores indicate higher levels of perceived stress. In this study, the total score was used for analysis.
  units on a scale | 25.35 (4.67) | 21.87 (5.89) | 23.61 (5.28)
The subscale Anxiety in Trauma Symptom Checklist for Children [Mean (Standard Deviation); unit: units on a scale] — The Trauma Symptom Checklist for Children (TSCC), Anxiety Subscale, measures trauma-related anxiety symptoms in children and adolescents. The subscale includes 9 items rated on a 4-point scale from 0 (never) to 3 (almost all the time). Total scores range from 0 to 27, with higher scores indicating more severe anxiety symptoms.
  units on a scale | 9.37 (4.98) | 6.31 (3.00) | 7.84 (3.99)
The subscale Depression in Trauma Symptom Checklist for Children [Mean (Standard Deviation); unit: units on a scale] — The Trauma Symptom Checklist for Children (TSCC), Depression Subscale, measures trauma-related depressive symptoms in children and adolescents. The subscale includes 9 items rated on a 4-point scale from 0 (never) to 3 (almost all the time). Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
  units on a scale | 10.05 (4.26) | 8.19 (3.10) | 9.12 (3.68)

OUTCOME MEASURES:

1. Primary Outcome: Perceived Stress Scale
Description: The 10-item Perceived Stress Scale (PSS-10) measures perceived stress related to unpredictability, uncontrollability, and overload in daily life. Each item is rated on a 5-point scale from 0 (never) to 4 (very often), yielding a total score ranging from 0 to 40. Higher scores indicate higher levels of perceived stress. In this study, the total score was used for analysis.
Time Frame: 8 weeks
Population: Difference is due to drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CFT Group Intervention | Control Group
Number analyzed (Participants) | 15 | 13
units on a scale | 22.73 (3.84) | 20.85 (5.83)

2. Primary Outcome: The Subscale Anxiety in Trauma Symptom Checklist for Children
Description: The Trauma Symptom Checklist for Children (TSCC), Anxiety Subscale, measures trauma-related anxiety symptoms in children and adolescents. The subscale includes 9 items rated on a 4-point scale from 0 (never) to 3 (almost all the time). Total scores range from 0 to 27, with higher scores indicating more severe anxiety symptoms.
Time Frame: 8- weeks
Population: Difference is due to drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CFT Group Intervention | Control Group
Number analyzed (Participants) | 15 | 13
units on a scale | 10.87 (4.96) | 6.15 (3.93)

3. Primary Outcome: The Subscale Depression in Trauma Symptom Checklist for Children
Description: The Trauma Symptom Checklist for Children (TSCC), Depression Subscale, measures trauma-related depressive symptoms in children and adolescents. The subscale includes 9 items rated on a 4-point scale from 0 (never) to 3 (almost all the time). Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Time Frame: 8 weeks
Population: Difference is due to drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CFT Group Intervention | Control Group
Number analyzed (Participants) | 15 | 13
units on a scale | 11.33 (3.64) | 7.31 (3.43)

ADVERSE EVENTS:
Time Frame: One week after intervention, 8 weeks after intervention started.
Description: Participants were instructed to report any adverse events during the intervention period to the research assistants or group leader. Adverse events were also assessed post-intervention with the question: "Did the CFT training help you to feel better?" with one of the response options being: "No, it seems to have made it worse."
Arm/Group | CFT Group Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

LIMITATIONS AND CAVEATS:
This study has several limitations. It was a pilot RCT feasibility study with a small sample size and preliminary efficacy results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT05448014/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT05448014/SAP_001.pdf